CLINICAL TRIAL: NCT03124966
Title: Accuracy of Hemoglobin Measurement for Various Rainbow Pulse Oximeter Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR19443-56044
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Noninvasive Hemoglobin Sensor (Experimental): All subjects are enrolled into the test group and all will receive the pulse oximeter sensor.
  Interventions: Device: Pulse Oximeter sensor

INTERVENTIONS:
Device: Pulse Oximeter sensor

SUMMARY:
In this study, the concentration of hemoglobin within the subject's blood will be reduced in a controlled manner by administering fluids intravenously. The accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparison to hemoglobin measurements from a laboratory analyzer.

ELIGIBILITY:
Study Site 1:

Inclusion Criteria:

* Has physical status between ASA 1 or 2
* Able to communicate in English

Exclusion Criteria:

* Pregnant or sexually active without birth control.
* Hemoglobin less than 11g/dL
* Known alcohol or drug abuse
* Skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection
* Nail polish
* Head injury with loss of consciousness within the last year
* Known neurological and psychiatric conditions.
* Known concurrent chronic usage of psychoactive or anti-convulsive drugs within the last 90 days, or use in the last 7 days (i.e. tricyclic antidepressants, MAO inhibitors, lithium, neuroleptics, anxiolytics or antipsychotics. Except SSRIs
* Subject has any medical condition which, in the judgement of the investigator, renders them inappropriate for participation in this study, such as Raynaud's syndrome
* Hypertension: Systolic BP >= 140 mmHg or Diastolic BP >= 90 mmHg
* Baseline heart rate <50 beats per minute

Study Site 2:

Inclusion Criteria:

* Male or female
* 18-35 years of age
* Physical status of ASA I or II
* Able to read and communicate in English
* Has signed written informed consent
* If female, non pregnant. If female subject is currently sexually active and not on birth control they must have a negative pregnancy test prior to study enrollment.

Exclusion Criteria

* Age less than 18 yrs and greater than 35 years
* Hemoglobin less than 12 g/dL
* ASA physical status of III, IV, or V
* Pregnant or sexually active without birth control
* Subject has known drug or alcohol abuse
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails.
* Subject has experienced a head injury with loss of consciousness within the last year
* Subject has known neurological and psychiatric disorder that interferes with the subjects level of consciousness
* Known or concurrent chronic usage of psychoactive or anticonvulsive drugs within the last 90 days, or any use in the last 7 day (i.e. tricyclic antidepressants, MAO inhibitors, lithium, neuroleptics, anxiolytics or antipsychotics, except SSRIs).
* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study, such as Raynauds Syndrome.
* Hypertension: Systolic BP >140 mmHg or Diastolic BP > 90 mmHg.
* Baseline heart rate < 50 bpm.
* Inability to tolerate sitting still or minimal movement for up to 90 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Masimo Clinical Lab, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Noninvasive Hemoglobin Sensor
Started | 118
Completed | 118
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Noninvasive Hemoglobin Sensor
Number analyzed (Participants) | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 118
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 118

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.
Time Frame: 1-3 hours
Measure: Number; unit: g/dL
Arm/Group | Noninvasive Hemoglobin Sensor
Number analyzed (Participants) | 118
g/dL | 0.96

ADVERSE EVENTS:
Arm/Group | Noninvasive Hemoglobin Sensor
All-Cause Mortality (participants affected / at risk) | 0/118
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less